CLINICAL TRIAL: NCT01719614
Title: A Phase I, Open-Label Study in Healthy Subjects to Explore the Potential for a Pharmacokinetic Interaction Between Steady-State Rilpivirine and a Single Dose Of Metformin
Brief Title: A Study to Explore Pharmacokinetic Interaction Between Rilpivirine and Metformin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100909; TMC278IFD1004 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Rilpivirine; Metformin; Pharmacokinetics
MeSH Terms: interventions — Metformin; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rilpivirine+Metformin (Experimental): All participants will receive study medications in two sessions in a fixed, sequential order as a session 1 (a single dose of metformin on Day 1) followed by washout period (period when no treatment is received) of 4 days and then session 2 (rilpivirine on Day 5 to Day 17 with a single dose of metformin on Day 15).
  Interventions: Drug: Metformin; Drug: Rilpivirine

INTERVENTIONS:
Drug: Metformin — Type=exact number, unit=mg, number=850, form=tablet, route=oral. Participants will receive single dose of metformin on Day 1 and Day 15.
Drug: Rilpivirine — Type=exact number, unit=mg, number=25, form=tablet route=oral. Participants will receive 1 tablet of rilpivirine from Day 5 to Day 17.

SUMMARY:
The purpose of the study is to evaluate the effect of steady-state (constant concentration of medication in the blood) rilpivirine on pharmacokinetics (how a single dose of metformin is absorbed in the body, distributed within the body, and removed from the body) of a single dose of metformin, over time, in healthy adult participants.

DETAILED DESCRIPTION:
This is a phase I, open-label (all people know the identity of the intervention) and sequential study (study medication is given in a sequence) in healthy participants, to investigate the pharmacokinetic interaction between steady-state rilpivirine and a single dose of metformin. The study consists of 3 phases including, the screening phase (28 days before enrollment), treatment phase (19 days), and the follow-up phase (7 days after the last intake of study medication). All participants will receive study medications in two sessions in a fixed, sequential order as a session 1 (a single dose of metformin on Day 1) followed by washout period (period when no treatment is received) of 4 days and then session 2 (rilpivirine on Day 5 to Day 17 with a single dose of metformin on Day 15). The duration of the study is approximately 54 days. Safety evaluations including adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination (including skin examination) will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy on the basis of physical examination, medical history, vital signs, electrocardiogram, the results of blood biochemistry and hematology tests and a urinalysis performed at screening
* Participant must have a Body Mass Index of 18.5 to 30.0 kg/m2
* Male participants should agree to protocol-defined use of effective contraception and women must be postmenopausal or surgically sterile
* Female participants must have a negative pregnancy test at screening
* Participants must be non-smoking for at least 3 months prior to screening

Exclusion Criteria:

* A positive Human immunodeficiency virus (HIV)-1 or HIV-2 test and Hepatitis A, B or C infection at screening
* Currently active clinically significant gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, endocrine, renal, hepatic, respiratory, inflammatory or infectious disease with any history of clinically significant skin disease
* Any history of tuberculosis, ocular herpes, or uveitis
* Have previously participated in more than one study with etravirine - TMC120 (dapivirine) and/or rilpivirine
* Participants with abnormal laboratory values at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma analyte concentration (Cmax) of metformin | Day 1 and Day 15
Actual sampling time to reach the maximum plasma analyte concentration (tmax) of metformin | Day 1 and Day 15
Area under curve from time of administration up to the last time point with a measurable plasma analyte concentration after dosing (AUClast) of metformin | Day 1 and Day 15
AUC extrapolated to infinity of metformin | Day 1 and Day 15
  AUC extrapolated to infinity, calculated as AUClast + Clast/apparent terminal elimination rate constant, where Clast is the last measurable plasma analyte concentration; extrapolations of more than 20 percent of the total AUC are reported as approximations.
Apparent terminal elimination rate constant of metformin | Day 1 and Day 15
  Apparent terminal elimination rate constant will be estimated by linear regression using the terminal log-linear phase of the logarithmic transformed conentration versus time data.
Apparent terminal elimination half-life of metformin | Day 1 and Day 15

SECONDARY OUTCOMES:
Predose plasma analyte concentration (C0h) of rilpivirine | Day 12, Day 13, Day 14, Day 15, Day 17, Day 18
Minimum observed plasma analyte concentration (Cmin) of rilpivirine | Day 15
Maximum observed plasma analyte concentration (Cmax) of rilpivirine | Day 15
Actual sampling time to reach the maximum plasma analyte concentration (tmax) of rilpivirine | Day 15
Observed plasma analyte concentration at the end of the 24-hour dosing interval (C24h) | Day 15
AUC from time of administration up to 24 hours after administration (AUC24h) | Day 15
Average steady-state plasma concentration (Css,av) | Day 15
  Css,av is calculated by AUC dosing interval/dosing interval at steady-state
Fluctuation index (FI) | Day 15
  FI, percentage fluctuation is variation between maximum and minimum plasma concentration at steady-state
Number of participants with adverse events as a measure of safety and tolerability | Up to 54 Days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Overland Park, Kansas, United States